CLINICAL TRIAL: NCT04573114
Title: Cerebral Hemodynamics During Early Verticalization After (Successful) Thrombectomy Poststroke
Acronym: CHEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01732
Record Dates: First submitted 2020-09-03; First posted 2020-10-05 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Stroke; Healthy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke subjects
  Interventions: Procedure: Verticalization
- Healthy
  Interventions: Procedure: Verticalization

INTERVENTIONS:
Procedure: Verticalization — Progressive levels of verticalization

SUMMARY:
This is a proof-of-concept study with a prospective observational design, where the association between progressive levels of verticalization and cerebral blood flow velocity (Ultrasound) in subacute stroke patients and healthy subjects will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic stroke in the territory of the middle cerebral artery (MCA)
* ≤12 hours after mechanical thrombectomy
* Conscious
* Hemodynamically stable
* 18 years or older
* Informed consent of the patient and/ or legal representative

Exclusion Criteria:

* Verticalization not allowed according to treating physician
* Known pre-stroke disease affecting cerebral blood flow
* Temporal bone windows insufficient to enable ultrasound penetration
* Intubation anticipated or occurred
* Venous thromboembolism
* Symptomatic intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: •First-ever ischemic stroke in the territory of the middle cerebral artery (MCA)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood flow velocity | within 12 hours post thrombectomy
  Cerebral blood flow velocity measured with transcranial doppler ultrasound

SECONDARY OUTCOMES:
Blood pressure | within 12 hours post thrombectomy
  Systolic and Diastolic pressure
Heart rate | within 12 hours post thrombectomy
  Number of contractions (beats) of the heart per minute
Oxygen saturation | within 12 hours post thrombectomy
  Relative measure of the concentration of oxygen in the blood
Impairment caused by a stroke | within 12 hours post thrombectomy
  National Institutes of Health Stroke Scale - NIHSS (Maximum score 42 - higher scores mean a worse outcome)
Neurological status | within 12 hours post thrombectomy
  Glasgow Coma Scale - GCS (Maximum score 15 - higher scores mean a better outcome)
Adverse events | within 12 hours post thrombectomy
  headache, focal edema, seizures, hemorrhagic transformation

OTHER OUTCOMES:
Reperfusion after thrombectomy | within 12 hours post thrombectomy
  modified Thrombolysis in Cerebral Infarction
Perfusion imaging | within 24 hours post thrombectomy
  Cerebral blood flow
Disability | 3 month post stroke
  modified Rankin Scale - mRS (maximum score 6 - higher scores mean a worse outcome)
Health-related quality | 3 month post stroke
  Patient-Reported Outcomes Measurement Information System® 29
Independence in gait | 3 month post stroke
  Functional Ambulation Categories (Maximum score 5 - higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Luft, MD, Study Chair — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deseoe J, Rottenberger Y, Pipping T, Schwarz A, Lehmann A, Veerbeek JM, Wegener S, Luft AR, Held JPO, Globas C. Very early tilt-table verticalization unmasks impaired cerebral autoregulation within 24 h after endovascular thrombectomy: a transcranial Doppler study. Front Neurol. 2026 Jan 6;16:1709991. doi: 10.3389/fneur.2025.1709991. eCollection 2025. PMID 41567543
- [Derived] Deseoe J, Schwarz A, Pipping T, Lehmann A, Veerbeek JM, Luft AR, Wegener S, Globas C, Held JPO. Cerebral blood flow velocity progressively decreases with increasing levels of verticalization in healthy adults. A cross-sectional study with an observational design. Front Neurol. 2023 Apr 17;14:1149673. doi: 10.3389/fneur.2023.1149673. eCollection 2023. PMID 37139076